CLINICAL TRIAL: NCT00513253
Title: Relative Bioavailability of Four Alternative Oral Formulations Versus the Current Tablet Formulation of Lapatinib
Brief Title: A Phase I Study to Test Alternate Oral Formulations vs the Current Tablet Formulation of Lapatinib
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: It was determined not to be needed based on the clinical development plan of Tykerb.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EGF101950
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Subjects
Keywords: lapatinib; Healthy Adult Volunteer
MeSH Terms: interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lapatinib

SUMMARY:
This study is designed to estimate the relative bioavailability of alternative lapatinib oral formulations compared to the current tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy as defined per protocol.
* The subject is male or female.

  * A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:
* Has had a documented (medical report verification) hysterectomy or double oophorectomy or
* Is 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy or
* Is post-menopausal (defined as females older than 45 years of age with 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels higher than 40 mIU/ml)

  * Childbearing potential, has a negative serum pregnancy test at Screening, and agrees to one of the following :
* Complete abstinence from sexual intercourse from two weeks prior to administration of the study drug and throughout the study, and through the follow-up visit which will occur within 10 to 14 days after completion of the last treatment.
* Vasectomized partner
* Intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm).
* Hormonal contraceptive plus male condom.
* Age: 18 to 60 years inclusive.
* BMI within the range 19 to 31.0 kg/m2.
* Able to swallow and retain oral medication.
* The subject is willing to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject is able to understand and comply with protocol requirements and instructions and is likely to complete the study as planned.
* A signed and dated written informed consent is obtained from the subject or the subject's legally acceptable representative prior to screening.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the Principal Investigator considers the subject unfit for the study.
* The subject meets ECG-related exclusion criteria listed in the protocol or has serum magnesium or potassium below the normal range at screening.
* The subject has a history of drug or other allergy, which, in the opinion of the Principal Investigator, contraindicates participation.
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, including but not limited to Tarceva (erlotinib) or Iressa (gefitinib).
* The subject has a history of sensitivity to heparin or heparin-induced thrombocytopenia (applicable if heparin is used during pharmacokinetic sampling).
* The subject participated in a study with a new molecular entity or any other trial during the previous 30 days.
* The subject donated blood in excess of 500 mL within 56 days prior to dosing or intends to donate in the month after completing the study.
* Use of prescription or non-prescription drugs (including vitamins and herbal supplements) within two weeks prior to dosing or during the study, however, acetaminophen up to two grams per day is acceptable.
* History of alcohol/drug abuse or dependence within 12 months of the study as per protocol.
* The subject is a smoker or has smoked in the last four months.
* The subject tested positive for hepatitis C antibody, hepatitis B surface antigen, or HIV antibody.
* The subject has a positive urine test for drugs of abuse or is positive for alcohol use at pre-study screening.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final PK blood sample.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Plasma levels for lapatinib will be done at: | Day 1, Day 2, Day 3 for each Treatment Period

SECONDARY OUTCOMES:
Medical History | at screening
Physical Exam | at screening & follow-up (f/u)
Continuous Adverse Event monitoring | throughout the study
Vital Signs, ECGs, & Lab tests | at screening, Day 1, and f/u
Response to questionnaire regarding taste and aesthetics of suspension formulations under evaluation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States